CLINICAL TRIAL: NCT00956670
Title: The LymphEdema and Gynecologic Cancer (LEG) Study: Incidence, Risk Factors, and Impact in Newly Diagnosed Patients
Brief Title: Lymphedema After Surgery in Patients With Endometrial Cancer, Cervical Cancer, or Vulvar Cancer
Acronym: LEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GOG-0244; NCI-2011-01932 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000646813; GOG-0244 (Other: NRG Oncology); GOG-0244 (Other: DCP); GOG-0244 (Other: CTEP); U10CA101165 (NIH); UG1CA189867 (NIH)
Record Dates: First submitted 2009-08-08; First posted 2009-08-11 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Lymphedema; Stage IA Cervical Cancer; Stage IA Uterine Corpus Cancer; Stage IA Vulvar Cancer; Stage IB Cervical Cancer; Stage IB Uterine Corpus Cancer; Stage IB Vulvar Cancer; Stage II Uterine Corpus Cancer; Stage II Vulvar Cancer; Stage IIA Cervical Cancer; Stage IIIA Vulvar Cancer; Stage IIIB Vulvar Cancer; Stage IIIC Vulvar Cancer; Stage IVB Vulvar Cancer
MeSH Terms: conditions — Lymphedema; Uterine Cervical Neoplasms; Vulvar Neoplasms

ARMS (1):
- Supportive care (lymphedema assessment) (Experimental): Patients with vulvar cancer undergo a radical vulvectomy or hemi-vulvectomy followed immediately by an ipsilateral or bilateral inguinal-femoral lymphadenectomy. (Closed to accrual as of June 9, 2014)
  Patients with cervical cancer undergo a radical hysterectomy or trachelectomy and bilateral pelvic lymphadenectomy +/- para-aortic nodal sampling via vaginal, laparoscopic, or open route.
  Patients with endometrial cancer undergo a laparoscopic-assisted vaginal hysterectomy, a total laparoscopic hysterectomy, or total abdominal hysterectomy with pelvic lymphadenectomy +/- para-aortic node sampling.
  Patients undergo limb measurements at baseline, weeks 4-6, and at 3, 6, 9, 12, 18, and 24 months.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Procedure: Study of High Risk Factors; Procedure: Therapeutic Conventional Surgery; Procedure: Therapeutic Laparoscopic Surgery; Procedure: Therapeutic Lymphadenectomy

INTERVENTIONS:
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Procedure: Study of High Risk Factors — Undergo lymphedema assessment
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Procedure: Therapeutic Laparoscopic Surgery — Undergo surgery
Procedure: Therapeutic Lymphadenectomy — Undergo lymphadenectomy

SUMMARY:
This clinical trial studies lymphedema after surgery in patients with endometrial cancer, cervical cancer, or vulvar cancer. Collecting information over time about how often lymphedema occurs in patients undergoing surgery and lymphadenectomy for endometrial cancer, cervical cancer, and vulvar cancer may help doctors learn more about the disease and plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To prospectively estimate the incidence of lower extremity lymphedema in patients undergoing radical surgery with a concurrent lymphadenectomy with a concurrent lymphadenectomy for a gynecologic malignancy.

II. To identify risk factors for the development of lower extremity lymphedema following radical surgery among patients with any one of the three types of gynecologic malignancy studied and to develop a corresponding predictive model.

SECONDARY OBJECTIVES:

I. To identify the effect that lower extremity lymphedema has on quality of life (QOL) (as measured with Functional Assessment of Cancer Therapy - General [FACT-G] + disease specific subscale), psychological adjustment (as measured with Impact of Events Scale [IES] and Functional Assessment of Chronic Illness Therapy [FACIT] body image items) and physical disability (of lower extremity as measured with Lower Extremity Functional Scale [LEFS]) and physical function(as measured by FACT-Functional Wellbeing [FW] subscale, FACIT disease specific items & patient-reported outcomes measurement information system [PROMIS] items) and to investigate potential protective mechanisms (FACT-Social Wellbeing [SW] subscale and patient characteristics).

II. To explore if patient self-reported symptoms (as measured with the lymphedema [LE] Symptom Measure [Cancer Lymphedema Questionnaire (GCLQ)]) are associated with the development of lymphedema in patients undergoing radical surgery for gynecologic malignancy.

TERTIARY OBJECTIVES:

I. To explore the effect of moderate or severe lymphedema (primary endpoint) on QOL outcomes, as measured by the FACT-General (G) questionnaire.

OUTLINE:

Patients with vulvar cancer undergo a radical vulvectomy or hemi-vulvectomy followed immediately by an ipsilateral or bilateral inguinal-femoral lymphadenectomy. (Closed to accrual as of June 9, 2014)

Patients with cervical cancer undergo a radical hysterectomy or trachelectomy and bilateral pelvic lymphadenectomy +/- para-aortic nodal sampling via vaginal, laparoscopic, or open route.

Patients with endometrial cancer undergo a laparoscopic-assisted vaginal hysterectomy, a total laparoscopic hysterectomy, or total abdominal hysterectomy with pelvic lymphadenectomy +/- para-aortic node sampling.

Patients undergo limb measurements at baseline, weeks 4-6, and at 3, 6, 9, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be registered into three distinct groupings, and each group will be analyzed as a separate study:

  * Patients who will undergo or have undergone hysterectomy/bilateral salpingo-oophorectomy (BSO) and pelvic lymphadenectomy +/- para-aortic node sampling via open or laparoscopic technique for clinical stage I-II or surgical stage I-III uterine carcinoma, including those receiving postoperative adjuvant therapy; patients enrolling after surgery may have a pathologic stage of I-III OR
  * Patients who will undergo or have undergone radical hysterectomy or trachelectomy and pelvic lymphadenectomy +/- para-aortic node sampling via open or laparoscopic technique for clinical stage IA-IIA cervical carcinoma, including those receiving postoperative adjuvant therapy OR
  * Patients with vulvar cancer who will undergo or have undergone definitive surgery for primary stage I-IV vulvar cancer who will or have received a radical vulvectomy or radical local excision with concurrent unilateral or bilateral inguinal or inguinal-femoral lymphadenectomy; patients who are going to receive multi-modality therapy (radiation +/-chemotherapy) after undergoing surgery are eligible; patients may undergo sentinel node mapping as long as it is followed by a full lymphadenectomy; (note: enrollment of vulvar patients was closed on June 9, 2014; no vulvar patients will be enrolled after closure of this arm)
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must have a serum albumin level of >= 3.0 within 14 days of entry
* Surgery must occur within 5 business days before study entry or within eight weeks after study entry

Exclusion Criteria:

* Patients with any prior clinical history of lower extremity lymphedema
* Patients who have a history of congestive heart failure, chronic renal disease, or chronic liver disease
* Patients with a prior history of chronic lower extremity swelling
* Patients with a Gynecologic Oncology Group (GOG) performance grade of 3 or 4
* Patients with a history of other invasive malignancies if their previous cancer treatment included any of the surgical procedures
* Patients who have had prior lower extremity vascular surgery (arterial or venous)
* Patients who have had prior pelvic, abdominal, inguinal, or lower extremity radiation therapy
* Patients who have had or are going to receive another elective surgery during the same operative event as their pelvic (cervical or uterine cancers) or inguinal (vulvar) lymphadenectomy
* Vulvar patients, from June 9, 2014 on
* Patients cannot be enrolled on the trial unless there is at least one person at the participating site who has been trained in performing limb measurements
* Patients who do not undergo or have not undergone the lymphadenectomy portion of the procedure
* Patients who enter the study and then undergo sentinel node biopsy without the intention of undergoing complete lymphadenectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1055 (Actual)
Dates: Start 2012-06; Primary Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Incidence of lymphedema, assessed through volumetric measurements using serial circumferential measurements performed from 10 cm above the heel to the inguinal crease at 10 cm intervals | Up to 24 months
  A competing risks analysis will be required to estimate the cumulative incidence of lymphedema. Transition probabilities in the Markov Chain will be estimated by simple proportions, ignoring covariates, to address this primary objective. Confidence intervals for the cumulative incidence of lymphedema then will be computed using the Delta Method, utilizing the fact that the transition proportions have and asymptotic multivariate normal distribution.
Risk factors for the development of lower extremity lymphoma in patients with endometrial cancers | Up to 24 months
  If risk factors are identified, a model will be developed to predict the level of risk (low, moderate, high) of lymphedema following gynecologic cancer treatment overall, and following treatment for endometrial cancer specifically. The predictive power of the models for these rates will be assessed.

SECONDARY OUTCOMES:
Patient self-reported symptoms | Up to 24 months
  Whether the patient self-reported symptoms are associated with the development of lymphedema wit be explored.
Quality of life | Up to 24 months
  As measured by the FACT QOL scale, psychological adjustment as measured by the Impact of Events Subscale (IES), and FACIT body image items, physical disability as measured by the Lower Extremity Functional Scale -(LEFS) and PROs of physical health status/function (sexual), as measured by FACT-FW; FACIT & PROMIS.
Risk factors for the development of lower extremity lymphoma in patients with cervical cancers | Up to 24 months
  If risk factors are identified, a model will be developed to predict the level of risk (low, moderate, high) of lymphedema following gynecologic cancer treatment overall, and following treatment for endometrial cancer specifically. The predictive power of the models for these rates will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Barakat, Principal Investigator — NRG Oncology
Locations (213):
- United States (213):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Gynecologic Oncology Group of Arizona, Phoenix, Arizona
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Carle on Vermilion, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Union Hospital of Cecil County, Elkton, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - New Hanover Regional Medical Center/Zimmer Cancer Center, Wilmington, North Carolina
  - Southeast Clinical Oncology Research (SCOR) Consortium NCORP, Winston-Salem, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming